CLINICAL TRIAL: NCT05228574
Title: Treatment of Vascular Stiffness in Patients With Autosomal Dominant Polycystic Kidney Disease
Brief Title: Treatment of Vascular Stiffness in ADPKD
Acronym: TRAMPOLINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, dr. M. Salih, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL72836.340.10
Record Dates: First submitted 2022-01-12; First posted 2022-02-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Autosomal Dominant Polycystic Kidney
Keywords: Polycystic kidney disease; Amiloride; Salt; Hypertension
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic Kidney Diseases; Hypertension | interventions — Sodium Chloride; Sodium Chloride, Dietary; Amiloride

STUDY DESIGN:
Intervention Model Description: This is a single-centre, randomized, double-blinded, and placebo-controlled clinical trial with a secondary open-label part.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-salt group (group 1) (Active Comparator): All participants will be subjected to a low-salt diet (3.5 grams/day) for six weeks.
  Group 1 will receive sodium chloride capsules (6 grams/day) for four weeks. In the last two weeks of the trial, all participants will be treated with amiloride tablets (20 mg daily) in open-label setting.
- Low-salt group (group 2) (Placebo Comparator): All participants will be subjected to a low-salt diet (3.5 grams/day) for six weeks.
  Group 2 will receive placebo capsules (6 grams/day) for four weeks. In the last two weeks of the trial, all participants will be treated with amiloride tablets (20 mg daily) in open-label setting.
  Interventions: Dietary Supplement: Placebo; Drug: Amiloride Hcl 5mg Tab

INTERVENTIONS:
Dietary Supplement: Sodium chloride (NaCl) — Sodium chloride capsules 6 grams per day for 4 weeks.
  Other Names: Table salt
Dietary Supplement: Placebo — Placebo capsules, 6 grams per day for 4 weeks.
  Arms: Low-salt group (group 2)
Drug: Amiloride Hcl 5mg Tab — Amiloride 5mg tablets, 20 mg per day for two weeks in open-label setting.
  Other Names: Amiloride
  Arms: Low-salt group (group 2)

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD) is the most common inherited kidney disease characterized by cystic kidneys and caused by mutations in the polycystic kidney disease and other rare genes. It is associated with salt-sensitive hypertension, which accounts for the majority of morbidity and mortality. About 70% of patients with ADPKD develop hypertension, prior to the onset of kidney function decline. Early onset hypertension, despite its treatment, is independently associated with rapid kidney function decline. The investigators hypothesize that a high-sodium diet in patients with ADPKD is required for the development of vascular stiffness, which precedes hypertension, and that treatment with amiloride reverses this phenomenon.

DETAILED DESCRIPTION:
Objective of the study:

The investigators aim to investigate if arterial stiffness is exacerbated due to a high-salt diet in patients with ADPKD. The investigators also aim to explore whether treatment with amiloride prevents the arterial stiffness caused by a high-salt diet.

Study design:

Randomized, double blinded and placebo-controlled clinical trial with open-label treatment with amiloride

Study population:

Adults with ADPKD with an estimated glomerular filtration rate (CKD-EPI) of ≥ 60 ml/min/1.73m2

Intervention:

All participants will be subjected to a low-salt diet (3,5 grams/day) throughout the study for a total of 6 weeks. After a run-in period of 2 weeks, participants will be randomized into two treatment groups:

Group 1: Sodium chloride capsules (6 grams/day) for 2 weeks, combined with amiloride (20 mg/day) in last 2 weeks Group 2: Placebo capsules for 2 weeks, combined with amiloride (20 mg/day) in last 2 weeks.

Primary study parameters/outcome of the study:

The three primary outcomes of this study are a difference in central arterial stiffness (pulse wave velocity, PWV) between:

1. The high-salt group versus low-salt group;
2. The high-salt group: before versus after amiloride treatment;
3. The low-salt group: before versus after amiloride treatment.

The burden of participation includes:

* A dietary salt restriction of 3.5 grams/day for a total period of 6 weeks
* Salt supplementation or placebo for a total period of 4 weeks
* Drug intervention with amiloride during the last 2 weeks
* Hospital visits

ELIGIBILITY:
Inclusion Criteria:

* Adults with typical ADPKD diagnosed based on Ravine criteria and/or a documented Pkd 1 or 2 mutation
* Chronic kidney disease epidemiology collaboration equation estimated glomerular filtration rate ≥60 ml/min/1.73m2
* Ability to provide informed consent

Exclusion Criteria:

* Uncontrolled hypertension, defined as an office blood pressure of ≥160/ ≥90 mmHg with or without antihypertensive treatment
* Concomitant use of ≥ 3 antihypertensive medications
* When antihypertensive treatment is prescribed for any other treatment indication than hypertension (e.g. cardia arrhythmia)
* Serum potassium levels >5.5 mmol/L (measured within last 6 months)
* History of liver disease (excluding liver cysts due to ADPKD)
* History of heart failure (cardiac ejection fraction < 35%) or cardiac arrhythmia
* History of diabetes mellitus
* Active infection or antibiotic therapy
* Immunosuppressive therapy within the last year
* Concomitant use of drugs that could influence blood pressure and/or disease progression (Tolvaptan/non-steroidal anti-inflammatory drugs (NSAIDs)/chemotherapy), excluding < 3 antihypertensive drugs
* Actual pregnancy or unwillingness to adhere to reproductive precautions during the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness induced by high salt diet | At week 3, week 5
  Difference in central arterial stiffness, measured as the pulse wave velocity (PWV), in high-salt group versus low-salt group.
Effect of treatment with amiloride on arterial stiffness in high-salt group | At week 5 and at week 7
  Difference in central arterial stiffness, measured as the pulse wave velocity (PWV), before versus after amiloride treatment in high-salt group.
Effect of treatment with amiloride on arterial stiffness in low-salt group | At week 5 and at week 7
  Difference in central arterial stiffness, measured as the pulse wave velocity (PWV), before versus after amiloride treatment in low-salt group.

SECONDARY OUTCOMES:
Blood pressure | At week 3, week 5 and at at week 7
  24-hours ambulatory blood pressure measurement (Mobil-O-Graph).
Salt tasting thresholds | At inclusion, week 3, week 5 and at week 7
  Sodium chloride (NaCl) solutions with different concentrations to assess the salt tasting thresholds.
Skin sodium accumulation | At week 3, week 5 and at week 7
  In a subgroup of participants, tissue sodium concentration (23Na) will be assessed noninvasively using a contrast-free 23 Na-MRI scan.
Markers of (vascular) inflammation and endothelial dysfunction | At inclusion, week 3, week 5 and at week 7
  Blood biomaterials will be collected at the visits. We will measure inflammatory markers including the high-sensitivity C-reactive protein, interleukin-6 and tumor necrosis factor-α, and other relevant markers for endothelial dysfunction including the adhesion molecules intercellular cell adhesion molecules-1, vascular cell adhesion molecules-1 and endothelin-1.

CONTACTS AND LOCATIONS:
Overall Officials: M. Salih, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus University Medical Centre Rotterdam, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039